CLINICAL TRIAL: NCT04931784
Title: Prospective, Open, Randomized Study Comparing the Effects of Ultimaster® Stents Treated With Conventional Methods on Coronary Artery Lesions Compared to the Most Dilated Coronary Vessels
Brief Title: Effect of Ultimaster Stents Treated to the Most Dilated Coronary Vessels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inha University Hospital (Other)
Collaborators: Terumo Corporation (Industry)
Responsible Party: Principal Investigator, Sang-Don Park, Associate Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INHAUH 2018-03-009
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Vasodilation; Coronary Artery Disease
MeSH Terms: conditions — Aneurysm; Coronary Artery Disease | interventions — Nitrates

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrate Group (Active Comparator): with administration of intra-coronary nitrate before percutaneous coronary intervention
  Interventions: Drug: Nitrate
- Control Group (Placebo Comparator): without administration of intra-coronary nitrate before percutaneous coronary intervention
  Interventions: Drug: Nitrate

INTERVENTIONS:
Drug: Nitrate — Administration of intra-coronary nitrate before percutaneous coronary intervention
  Other Names: No intervention

SUMMARY:
In patients with vasospasm or with negative remodeling, various vasodilator drugs used during coronary angiography can dilate the diameter of the reference vessel to measure the exact vessel size. In particular, nitrates are well known to induce pharmacological vasodilatory effects through vascular smooth muscle relaxation In actual clinical practice, it has been reported that when oral or spray-type nitrate preparations are administered to coronary artery stenosis lesions, the diameter of the reference vessel expands by about 10% compared to the existing vessel diameter. This may enable larger stenting in coronary artery stenosis lesions. Although many patients with vascular stenosis are accompanied by vasospasm and voice remodeling, in actual clinical practice, administration of vasodilators is only used in a small number of patients at the discretion of the surgeon. Nitrate vasodilators administered during coronary angiography are low-dose and short-acting drugs, and although a small number of patients may experience side effects such as short-term lowering of blood pressure, no serious side effects are reported .

On this background, this study is to evaluate whether there is a difference in the diameter of the Ultimaster® stent treated with the conventional method compared to the maximally dilated coronary artery, and to evaluate the stability and effectiveness after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years old
* evidence of coronary artery disease including asymptomatic ischemia stable angina acute coronary syndrome (unstable angina, non-ST segment elevation

  * myocardial infarction, ST segment elevation myocardial infarction).
* coronary artery diameter 2.25~3.5mm, stenosis 50% or more
* Those who voluntarily agreed in writing to participate in this clinical study

Exclusion Criteria:

* instability or psychogenic shock within 24 hours before percutaneous coronary intervention
* life expectancy no longer than 1 year
* hypersensitivity or contraindications to the following drugs or substances: heparin, aspirin, clopidogrel
* patients whom researchers think unsuitable for participation in this study

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean stent diameter | Immediately after percutaneous coronary intervention

SECONDARY OUTCOMES:
Failure rate of target lesion for 1-year (combination of cardiac death, target vascular myocardial infarction, target vascular revascularization) | 1 year after percutaneous coronary intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon GS, Choi SH, Kwon SW, Park SD, Woo SI. A prospective double-blinded randomized study on drug-eluting stent implantation into nitrate-induced maximally dilated vessels in patients with coronary artery disease. Trials. 2023 Jul 18;24(1):460. doi: 10.1186/s13063-023-07497-5. PMID 37464355